CLINICAL TRIAL: NCT03711734
Title: Feasibility of Electro Auricular Acupuncture for Analgesia After ACL Surgery: The Feasibility of Patient Blinding and Effects on Early Postoperative Pain
Brief Title: Acupuncture ACL (Anterior Cruciate Ligament)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2018-1478
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: ACL; ACL Injury; Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Rupture; Anesthesia
Keywords: Acupuncture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture + Standard of Care (Experimental): Patients will receive spinal anesthesia (4 cc Mepivacaine) with IV sedation. Intraoperative anti-emetics will consist of IV odansetron and IV dexamethasone. Intra-operative analgesics will include IV Ketamine, IV Ketorolac, and IV Acetaminophen.
  Patients will have ATP acupuncture (8 ear points - Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) bilaterally with electrostimulation at Shen men and Hypothalamus at 30 hz.
  Interventions: Other: Acupuncture + Standard of Care
- No acupuncture + Standard of Care (No Intervention): Patients will receive spinal anesthesia (4 cc Mepivacaine) with IV sedation. Intraoperative anti-emetics will consist of IV odansetron and IV dexamethasone. Intra-operative analgesics will include IV Ketamine, IV Ketorolac, and IV Acetaminophen.
  Patients will not have ATP acupuncture (8 ear points - Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) bilaterally.

INTERVENTIONS:
Other: Acupuncture + Standard of Care — Acupuncture is a nonpharmacologic pain management modality that has been shown to provide superior analgesia for acute pain. This will be combined with our facility's standard of care anesthesia and pain management plan.
  Arms: Acupuncture + Standard of Care

SUMMARY:
Acupuncture research in regards to PONV has been fairly well established, however, studies about perioperative pain control and acupuncture are a little more murky. In 2008, a meta analysis looked at randomized controlled studies and found that while acupuncture was shown to decrease pain, there were limitations including credible placebo or sham intervention, and thus, blinding. The main purpose of this feasibility trial is to determine whether or not adequate blinding is possible in the intraoperative setting with the patient sedated.

DETAILED DESCRIPTION:
According to the most recent survey conducted by the national center for complementary and integrative health (a branch of the National Institutes of Health) in 2007, the use of complementary alternative medicine (CAM) has increased significantly from 2002 (the previous survey). In the 2007 survey, in the United States alone, 38% percent of adults and 12% of children use some form of CAM. It has been 10 years since that survey report, there is little doubt that these numbers have only increased. According to the National Center for Health Statistics on the expenditures on CAM in 2012 - for just adults utilizing specialists, such as acupuncturists, $14.1 Billion was spent. With this increasing demand of such treatment modalities by patients, conventional practitioners will need to be, at the very least, well versed enough to recommend for or against these modalities. In addition, the current opioid epidemic is on the forefront of the public mind. Recently declared a public health emergency by the President, alternative means of postoperative pain control is a necessity and integrative medicine is a low cost, safe, and effective adjuvant/alternative

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACL Surgery with a participating surgeon
* English Speaking
* Patients at least 12 years old
* Planned spinal anesthesia without peripheral nerve block (rescue block is okay)

Exclusion Criteria:

* Patients under the age of 12
* Non-English speaking patients
* Patients planning on having general anesthesia
* Planned preop peripheral nerve block
* Patients with the inability to understand/follow study protocol
* Patients with pacemaker/AICD
* Non-native Ear/Previous scarring/surgical manipulation of ear
* Patients with contraindications to intra-op protocol
* Chronic pain patients
* Patients who have regularly used opioids for more than 6 weeks prior to surgery
* Patients with guages in their ears
* Patients who refuse to remove earrings/piercings prior to surgery
* Patients with nickel allergies (needles are made of nickel)

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cheng, MD, Principal Investigator — Hospital for Special Surgey
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng SI, Norman RM, DeMeo D, Zhong H, Turteltaub LH, McCarthy MM, Marx RG, Strickland SM, Kelly AM. The Feasibility of Blinding Intraoperative Electro-Auricular Acupuncture Under Neuraxial Anesthesia. Med Acupunct. 2021 Aug 1;33(4):286-294. doi: 10.1089/acu.2021.0003. Epub 2021 Aug 17. PMID 34471447

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture + Standard of Care: Patients will receive spinal anesthesia (4 cc Mepivacaine) with IV sedation. Intraoperative anti-emetics will consist of IV odansetron and IV dexamethasone. Intra-operative analgesics will include IV Ketamine, IV Ketorolac, and IV Acetaminophen.
  Patients will have ATP acupuncture (8 ear points - Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) bilaterally with electrostimulation at Shen men and Hypothalamus at 30 hz.
  Acupuncture + Standard of Care: Acupuncture is a nonpharmacologic pain management modality that has been shown to provide superior analgesia for acute pain. This will be combined with our facility's standard of care anesthesia and pain management plan.
Period: Overall Study
Arm/Group | Acupuncture + Standard of Care | No Acupuncture + Standard of Care
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of all participants for whom baseline characteristics were measured, in each arm/group and in the entire study population (total)
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture + Standard of Care | No Acupuncture + Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11.1) | 29.8 (13) | 32 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Bang Blinding Index (BI)
Description: Patients' ability to determine whether or not they received acupuncture. The success of patient blinding in each group will be quantified using Bang Blinding Index (BI) which ranges from min = -1 to max = 1. Scores closest to 0 indicate a less likelihood that patients were able to guess which group they were randomized into. A score of 1 or -1 means that patients were able to guess which group they were in. This value is obtained by asking patients which group they believe they were randomly assigned to.
Time Frame: postoperative day 1
Population: One patient was lost to follow up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture + Standard of Care | No Acupuncture + Standard of Care
Number analyzed (Participants) | 20 | 19
score on a scale | 0.2 [-0.02 to 0.42] | 0.11 [-0.10 to 0.31]

2. Secondary Outcome: Numeric Rating Scale (NRS) Pain at Rest Scores
Description: Numeric Rating Scale (NRS) pain at rest on a scale of 0 (no pain) to 10 (worst pain ever imaginable). A lower score is a better outcome.
Time Frame: postoperative day 1
Population: One patient was lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture + Standard of Care | No Acupuncture + Standard of Care
Number analyzed (Participants) | 20 | 19
score on a scale | 4.3 (1.8) | 4.1 (1.9)

3. Secondary Outcome: Numeric Rating Scale (NRS) Pain With Movement Scores
Description: Numeric Rating Scale (NRS) pain with movement on a scale of 0 (no pain) to 10 (worst pain imaginable). A lower score is a better outcome.
Time Frame: postoperative day 1
Population: Some patients were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture + Standard of Care | No Acupuncture + Standard of Care
Number analyzed (Participants) | 19 | 18
score on a scale | 5.2 (1.9) | 4.6 (1.9)

4. Secondary Outcome: Opioid Consumption
Description: Measured in cumulative oral morphine equivalent. Each patient measured individually and then all patients' measurement was averaged.
Time Frame: day of surgery through postoperative day 1
Measure: Mean (Standard Deviation); unit: oral morphine equivalent
Arm/Group | Acupuncture + Standard of Care | No Acupuncture + Standard of Care
Number analyzed (Participants) | 20 | 20
oral morphine equivalent | 47.8 (34.6) | 46.3 (25.3)

ADVERSE EVENTS:
Time Frame: From when the patient is enrolled in the study (i.e., sign the consent form) to the last follow up contact with the patient (up to 1 year)
Description: Assessed across all 40 participants, 20 participants in each arm/group.
  No patients died or experienced an adverse event
Arm/Group | Acupuncture + Standard of Care | No Acupuncture + Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03711734/Prot_SAP_000.pdf